CLINICAL TRIAL: NCT07392112
Title: The Effect of Nada Yoga Music Therapy on Perceived Pain and Anxiety During the Labor Process
Brief Title: Nada Yoga Music Therapy for Pain and Anxiety in Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sinop University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SİNOPU-SİBEL1
Record Dates: First submitted 2026-01-01; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Labor Pain; Yoga; Music Therapy
Keywords: Labor pain; Anxiety; Nada Yoga music therapy
MeSH Terms: conditions — Labor Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This study is designed as a randomized controlled trial.
Who Masked: Participant
Masking Description: Due to the nature of the intervention (audible music), participants and healthcare providers could not be blinded to group allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nada Yoga music therapy (Experimental): Intervention Applied to the Intervention Group
  This intervention is a behavioral intervention. Participants in the experimental arm receiPregnant women in the intervention group will receive Nada Yoga music therapy after admission to the delivery room. The intervention will be implemented as follows:
  Selected music: A playlist consisting of special melodies, mantras, and nature sounds compatible with the philosophy of Nada Yoga, which have been proven to have a relaxing effect on brain waves, will be used.
  Duration of application: Music therapy will continue from the time of admission to the delivery room until birth occurs.
  Method of application: During this period, the pregnant women will listen to the music through speakers placed in the labor room.Pregnant women in the intervention group will listen to Nada Yoga music via speakers throughout labor after admission to the delivery room, and their pain and anxiety levels will be assessed using the VAS and the State Anxiety Inventory.
  Interventions: Other: Nada Yoga music therapy
- Control Group (No Intervention): Procedure Applied to the Control Group Pregnant women in the control group will not receive any music therapy, and standard obstetric care procedures will be followed. This group will be monitored throughout the labor process without any additional relaxing music or sound interventions.Pregnant women in the control group will receive only routine obstetric care throughout labor, without any music or additional relaxing interventions, and their pain and anxiety levels will be assessed using the VAS and the State Anxiety Inventory.

INTERVENTIONS:
Other: Nada Yoga music therapy — Nada Yoga music therapy
  Arms: Nada Yoga music therapy

SUMMARY:
This study was designed as a randomized controlled trial. Based on the power analysis (Cohen's d = 0.80, α = 0.05, power = 80%), a total of 52 pregnant women were included, with 26 participants in the intervention group and 26 in the control group. Pregnant women who met the inclusion criteria and provided written informed consent were randomly assigned to the groups using a computer-generated randomization method.

The intervention group received Nada Yoga music therapy after admission to the delivery room, and the intervention was continued until birth. The therapy consisted of music compatible with the philosophy of Nada Yoga, including relaxing melodies, mantras, and nature sounds, which were delivered via speakers placed in the labor room. The control group received standard obstetric care.

Data were collected using the Pregnant Woman Information Form, Labor Follow-up Form, Visual Analog Scale (VAS), and the Spielberger State Anxiety Inventory.

DETAILED DESCRIPTION:
This study was conducted as a randomized controlled trial. The sample size was determined through a power analysis based on an effect size of 0.80 (Cohen's d) obtained from a reference study, a significance level of 5% (α = 0.05), and a statistical power of 80% (1 - β = 0.80). The calculation for two independent groups indicated that a total of 52 pregnant women, with 26 participants in each group (26 in the intervention group and 26 in the control group), were required, and the study was completed with this sample size.

The study was carried out on two independent groups to evaluate the effectiveness of music therapy during the labor process. The intervention group consisted of pregnant women who received Nada Yoga music therapy, while the control group comprised pregnant women who received standard obstetric care. Pregnant women who met the inclusion criteria and voluntarily agreed to participate provided both verbal and written informed consent, after which they were randomly assigned to the intervention or control groups using a computer-generated randomization method.

Pregnant women in the intervention group received Nada Yoga music therapy after admission to the delivery room. As part of the intervention, a specially selected music playlist consistent with the philosophy of Nada Yoga-including relaxing melodies, mantras, and nature sounds known for their calming effects-was used. The music was delivered through speakers placed in the delivery room, and the intervention was continued uninterrupted from admission until birth. No music therapy was applied to the control group; these participants were followed throughout the labor process solely according to routine obstetric care protocols.

During the implementation of the study, pregnant women admitted to the labor clinic were informed about the aim, scope, and procedures of the research. Prior to the intervention, when cervical dilation reached 4-5 cm, data were collected from both groups using the Pregnant Woman Information Form, the Labor Follow-up Form, the Visual Analog Scale (VAS) for pain assessment, and the Spielberger State Anxiety Inventory.

Following the intervention, data collection was repeated in both groups at different stages of labor. Measurements were conducted during the active phase (cervical dilation of 4-7 cm) and the transition phase (cervical dilation of 8-10 cm). At these stages, the Pregnant Woman Information Form, the Labor Follow-up Form, the Visual Analog Scale (VAS), and the Spielberger State Anxiety Inventory were re-administered to assess pain and anxiety levels.

ELIGIBILITY:
Inclusion Criteria:

* Having no impairment in communication skills
* Voluntarily agreeing to participate in the study
* Being between 37-42 weeks of gestation
* Planning a vaginal delivery
* Having no high-risk factors during pregnancy
* Having a singleton pregnancy
* Having a vertex fetal presentation

Exclusion Criteria:

* Individuals with communication problems
* Those who do not volunteer to participate in the study
* Pregnant women before 37 weeks of gestation or after 42 weeks of gestation
* Pregnant women with a planned cesarean delivery
* Pregnant women with gestational diabetes, preeclampsia, or other obstetric risk factors
* Those with multiple pregnancies
* Those with non-vertex fetal presentations (e.g., breech, transverse)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant woman
Enrollment: 52 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measure | Before the intervention (when cervical dilatation reached 4-5 cm) and after the intervention during the active (4-7 cm) and transition (8-10 cm) phases of labor
  Before the intervention, when cervical dilatation reached 4-5 cm, the following assessments were conducted in pregnant women in both groups: collection of demographic and obstetric characteristics using the Personal Information Form and Labor Follow-up Form, assessment of pain intensity using the Visual Analog Scale (VAS), and measurement of anxiety levels using the Spielberger State Anxiety Inventory.

SECONDARY OUTCOMES:
Secondary Outcome Measure | Before the intervention (at 4-5 cm cervical dilatation) and after the intervention during the active (4-7 cm) and transition (8-10 cm) phases of labor
  After the intervention, assessments were conducted in both groups during different stages of labor: the active phase (4-7 cm cervical dilatation) and the transition phase (8-10 cm cervical dilatation) VAS This scale, which can be used horizontally or vertically, consists of a 10 cm line. It begins with "No pain" and ends with "Worst possible pain." Participants are asked to mark a point on the scale between 0 and 10 that best represents the pain they perceive Spielberger State Anxiety Inventory It is a self-report instrument consisting of short statements. The inventory is designed to assess an individual's anx.Scores obtained from the State Anxiety Scale theoretically range from 20 to 80. Scores below 36 indicate no anxiety, scores between 37 and 42 indicate mild anxiety, and scores of 42 and above indicate high anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Sibel YÜCETÜRK, pHd, Study Chair — SinopUniversity
Locations (2):
- Turkey (Türkiye) (2):
  - Sinop University, Sinop, Sinop
  - sinop University, Sinop, Sinop University

IPD SHARING:
Plan to Share IPD: No
Individual patient data obtained in this study will not be shared with other researchers in order to protect the privacy and confidentiality of the participants.

REFERENCES:
- [Result] Misto, R. (2016). Yoga of Sound music therapy system: techniques acting on autonomic nervous system. Nordic Journal of Music Therapy. https://doi.org/10.1080/08098131.2016.1180115. Misto, R. (2020). Therapeutic Musical Scales: Theory and Practice. , 6, 1-1. https://doi.org/10.21926/OBM.ICM.2102019. Singh, P. (2021). Exploring Current Music Therapy Practices in India. Voices: A World Forum for Music Therapy. https://doi.org/10.15845/voices.v21i3.3246. Sundar, S. (2005). Can Traditional Healing Systems Integrate With Music Therapy -